CLINICAL TRIAL: NCT01207986
Title: Early Lung Cancer Diagnosis in HIV Infected Population With an Important Smoking History With Low Dose CT: a Pilot Study
Acronym: EP48 HIV CHEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AO 781-38
Record Dates: First submitted 2010-09-16; First posted 2010-09-23 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Hiv Infection; Lung Cancer
MeSH Terms: conditions — HIV Infections; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT screening (Other): CT interpretations and lung biopsies are guided by a suggested workup algorithm, which is not imposed in each HIV-caring centre
  Interventions: Radiation: Low dose computed tomography (CT)

INTERVENTIONS:
Radiation: Low dose computed tomography (CT)

SUMMARY:
Early Lung Cancer diagnosis in a HIV-infected population with an important smoking history with low-dose CT: a pilot study: the HIV-CHEST study Objectives The main objective of this study is to evaluate the prevalence of lung cancers detected by low-dose computed tomography (CT) in a HIV-infected population with an important smoking history. Other objectives are (1) the evaluation of the types of lung cancers in this population, as well as (2) the staging of non small cell lung cancers, (3) the description of risk factors for all lung cancers, if they are numerous enough, and (4) the number of complications of diagnosis procedures during the study.

DETAILED DESCRIPTION:
Background Epidemiological studies in France and in the western world have shown that lung cancers are the first cause of mortality amongst the non-AIDS classifying cancers in HIV-infected individuals, despite the introduction of combination antiretroviral therapies. Compared to the general population, there is an increased risk of lung cancer in HIV-infected individuals, even after adjustment on smoking and age, estimated to be around 2.6 compared to the general population. Outcomes are dismal, as diagnoses in HIV-infected individuals are usually made at very advanced stages (usually stage III or IV) without screening. Two non-randomized studies of CT-screening in a non HIV-infected population exposed to smoking have shown an important rate of early lung cancer detection and a high level of survival at 5 or 10 years. Despite a probable high prevalence of lung cancer in the HIV-infected population, no lung cancer screening or early diagnosis studies have been realised, and the prevalence is yet to be determined. We deduced from different studies of non HIV-infected populations a 3% prevalence in the HIV-infected population.

Methods Prospective multicentric and national study evaluating the prevalence of lung cancers through low-dose CT of 450 individuals with a known HIV-infection, with a nadir level of TCD4 cells < 350/µl, ≥ 40 years old and with a smoking history ≥ 20 packs a year (either active or with <3 years of weaning). CT interpretations and lung biopsies are guided by a suggested workup algorithm, which is not imposed in each HIV-caring centre.

Inclusion and follow up period Inclusion period will be 9 months, followed, in case of the discovery of a small nodule, by a CT follow up scheme of up to two years from first diagnosis. The study closes after 26 months of follow up.

Awaited results For the first time, this prospective study of lung cancers will estimate the prevalence of these cancers screened in the HIV-infected population. Risks associated with the incidence of this cancer will be investigated, including potential immune factors. An increased number of stage I non small cell lung cancers are expected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* able to give written consent
* HIV positive serology
* Covered by French Social Security
* Nadir L TCD4 < 350/µl
* Rate of LTCD4 > 100/µl at inclusion
* Addiction to smoking > 20 packages years, active person or deprived since < 3 years

Exclusion Criteria:

* patients who suffered from comorbidity
* unaffiliated to the social healthy security french system
* Presence of an evolutionary cancer
* any evolutionary pathology classifying AIDS
* Pregnancy
* Recent lung infection (< 2 months)
* Be under protection (saving) of justice

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
the prevalence of lung cancers detected by lowdose computed tomography | Month 0

SECONDARY OUTCOMES:
the types of lung cancers in this population, | Month 1 Month 3 Month 12 Month 24 Month 26
the staging of non small cell lung cancers, | Month 1 Month 3 Month 12 Month 24 Month 26
description of risk factors for all lung cancers, | Month 1 Month 3 Month 12 Month 24 Month 26
number of complications of diagnosis procedures during study | Month 1 Month 3 Month 12 Month 24 Month 26

CONTACTS AND LOCATIONS:
Overall Officials: Alain Makinson, Principal Investigator — University Hospital, Montpellier; Antoine Cheret, Principal Investigator — CHU Tourcoing; Sophie Abgrall, Principal Investigator — Hospital Avicenne; Pierre Delamonicca, Principal Investigator — CHU NICE; Pierre Tattevin, Principal Investigator — Pontchaillou; Isabelle Poizot Martin, Principal Investigator — St Marguerite Marseille; Francois Raffi, Principal Investigator — Hotel Dieu Nantes; Claudine Duvivier, Principal Investigator — Necker Paris; David Zucman, Principal Investigator — Foch Suresnes; Jean Louis Couderc, Principal Investigator — Foch Suresnes; Tristan Ferry, Principal Investigator — La Croix Rousse Lyon; Jean Marc Mauboussin, Principal Investigator — Nîmes, CH Caremeau
Locations (1):
- Makinson, Montpellier, France

REFERENCES:
- See also: Related Info — http://anrs.fr